CLINICAL TRIAL: NCT06568133
Title: An Open-label, Multiple-dosing, Two-arms, One-sequence Study to Evaluate the Safety and Pharmacokinetics After Co-administration of UIC201603 and UIC201604 in Healthy Volunteers
Brief Title: Drug-drug Interaction Study Between UIC201603, and UIC201604
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea United Pharm. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: KUP-UI022-101
Record Dates: First submitted 2024-07-23; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2018-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): UIC201603 and co-administration of UIC201603 and UIC201604
  Interventions: Drug: UIC201603 and co-administration of UIC201603 and UIC201604
- Treatment B (Experimental): UIC201604 and co-administration of UIC201603 and UIC201604
  Interventions: Drug: UIC201604 and co-administration of UIC201603 and UIC201604

INTERVENTIONS:
Drug: UIC201603 and co-administration of UIC201603 and UIC201604 — * UIC201603 2 Caps/day for 7 days
  * Wash out 7 days
  * UIC201603 2 Caps/day + UIC201604 1 Tabs/day for 7 days
  Arms: Treatment A
Drug: UIC201604 and co-administration of UIC201603 and UIC201604 — * UIC201604 1 Tabs/day for 7 days
  * Wash out 7 days
  * UIC201603 2 Caps/day + UIC201604 1 Tabs/day for 7 daysadministration of UIC201603 and UIC201604
  Arms: Treatment B

SUMMARY:
An open-label, multiple-dosing, two-arms, one-sequence study to evaluate the safety and pharmacokinetics after co-administration of UIC201603 and UIC201604 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Subjects whose body weight over 55 kg and ranged ± 20% of calculated Ideal Body Weight;
2. Subjects without congenital disease, chronic disease, symptom or any clinical significance of a physical examination and questionnaires;
3. Subjects judged as healthy by laboratory tests including blood haematology, biochemistry, urinalysis and serologic tests;
4. Subjects able to read and understand a written informed consent, and willing to participate in the study.
5. For women, those who are confirmed not to be pregnant during a health examination

Exclusion Criteria:

1. Clinically significant, liver, kidney, nervous system, respiratory system, blood/tumor, urinary system, Mental disorders, especially cardiovascular diseases (e.g. hypertension, angina pectoris, heart failure, myocardial infarction, etc.) Those who have or have a history of diseases related to the endocrine system (diabetes, hyperlipidemia, etc.)
2. Bleeding (hemophilia, capillary fragility, intracranial hemorrhage, upper digestive tract hemorrhage, urinary tract hemorrhage, hemoptysis, vitreous hemorrhage, etc.) or such predispositions (active peptic ulcer, hemorrhagic stroke within the past 6 months, surgery within the past 3 months, proliferative diabetic retinopathy, uncontrolled Patients with high blood pressure)
3. Patients with atrial or ventricular displacement, patients with atrial fibrillation or flutter, ventricular tachycardia, ventricular fibrillation, or Patients with multifocal ventricular ectopic beats and patients with prolonged QT interval
4. Gastrointestinal diseases that may affect the absorption of investigational drugs (Crohn's disease, ulcers) acute or chronic pancreatitis, etc.) or gastrointestinal surgery (however, simple appendectomy or Those with a history of hernia surgery (excluding hernia surgery)
5. Those with a history of hypersensitivity to Cilostazol or other antiplatelet agents,
6. Same series as rosuvastatin, atorvastatain, simvastatin, etc. (HMG-CoA Hypersensitivity reaction to the components of reductase inhibitor or clinically significant Those with a history of hypersensitivity reaction
7. Galactose intolerance, Lapp lactase deficiency lactose deficiency or glucose-galactose malabsorption People with genetic problems such as malabsorption
8. If PT and aPTT are outside the allowable range (diagnostic laboratory reference values are 11-15 sec, respectively, 22.4-40.4 sec)
9. Vital signs show systolic blood pressure ≥ 140 mmHg or < 90 mmHg, diastolic blood pressure ≥ 95 Either mmHg or <60 mmHg, pulse rate ≥100 beats/min. Those who showed included figures
10. Those with high-density lipoprotein (HDL-cholesterol) less than 35 mg/dL
11. Those whose serum potassium concentration is less than 3.4 mEq/L or more than 5.5 mEq/L
12. Have a history of muscle disease or a personal or family history of hereditary muscle abnormalities ruler
13. Patients with biliary obstructive disease
14. Unexplained persistent elevation of serum transaminases or three times the upper limit of normal Patients with active liver disease including excess serum transaminase elevations
15. Patients with severe renal impairment (creatinine clearance calculated by the Cockcroft-Gault equation is 30 Those with less than mL/min)
16. Those with a history of drug abuse or a positive drug abuse test
17. Induction of drug metabolizing enzymes such as barbiturates within 1 month before the first administration date and Those who take suppressive drugs or drink excessively
18. Those who have taken any prescription medicine or herbal medicine within 2 weeks before the first medication date, or any over-the-counter medicine (OTC medicine) or vitamin supplement within 10 days (except, Depending on the investigator's judgment, you may participate in the clinical trial if other conditions are reasonable. has exist)
19. Participating in another clinical trial or bioequivalence test within 3 months before the first administration date Person who administered clinical trial drug
20. Donate whole blood within 2 months or component blood within 1 month before the first dose. or received a blood transfusion within 1 month before the first dose
21. For women, pregnant/nursing or currently using a medically acceptable form of contraception. Those who are not using contraception or are unable to maintain contraception during the clinical trial period
22. Clinical test performance The investigator may not conduct a clinical trial due to test results or other reasons. Those judged unsuitable for participation

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics(AUCss,τ) of Cilostazol and Active metabolites(OPC-13015, OPC-13213) | Day 7 and Day 21: -72, -48, -24, 0h, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24h
  Area under the serum drug concentration-time curve within a dosing interval at steady state
Plasma pharmacokinetics(Css,max) of Cilostazol and Active metabolites(OPC-13015, OPC-13213) | Day 7 and Day 21: -72, -48, -24, 0h, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24h
  Maximum concentration of drug in serum at steady state
Plasma pharmacokinetics(AUCss,τ) of Rosuvastatin | Day 7 and Day 21: -72, -48, -24, 0h, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24h
  Area under the serum drug concentration-time curve within a dosing interval at steady state
Plasma pharmacokinetics(Css,max) of Rosuvastatin | Day 7 and Day 21: -72, -48, -24, 0h, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24h
  Maximum concentration of drug in serum at steady state

CONTACTS AND LOCATIONS:
Overall Officials: Janghee Hong, M.D.,Ph.D, Principal Investigator — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim DH, Hong JH, Jung WT, Nam KY, Roh JS, Lee HJ, Moon J, Kim KY, Jung JG, Sunwoo J. Pharmacokinetic Drug-Drug Interaction between Cilostazol and Rosuvastatin in Healthy Participants. Am J Cardiovasc Drugs. 2025 Mar;25(2):267-276. doi: 10.1007/s40256-024-00686-w. Epub 2024 Nov 2. PMID 39487337